CLINICAL TRIAL: NCT06008756
Title: Phase 3 Randomized, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of MK-0616 in Reducing Major Adverse Cardiovascular Events in Participants at High Cardiovascular Risk
Brief Title: Enlicitide Decanoate (MK-0616 Oral PCSK9 Inhibitor) Cardiovascular Outcomes Study (MK-0616-015) CORALreef Outcomes
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0616-015; jRCT2071230064 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2022-502781-24-00 (Registry Identifier: EU CT); U1111-1285-4245 (Registry Identifier: UTN)
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Arteriosclerosis; Hypercholesterolaemia
MeSH Terms: conditions — Arteriosclerosis; Hypercholesterolemia | interventions — MK-0616

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enlicitide Decanoate (Experimental): Participants receive enlicitide decanoate 20 mg once daily.
  Interventions: Drug: Enlicitide Decanoate
- Placebo (Placebo Comparator): Participants receive placebo once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enlicitide Decanoate — Enlicitide Decanoate 20 mg tablet taken by mouth.
  Other Names: MK-0616
  Arms: Enlicitide Decanoate
Drug: Placebo — Placebo tablet matched to enlicitide decanoate taken by mouth.
  Arms: Placebo

SUMMARY:
This is a phase 3, randomized, placebo-controlled study of the efficacy and safety of enlicitide decanoate, an oral proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor, in participants with high cardiovascular risk. The primary objective is to evaluate the efficacy of enlicitide decanoate compared with placebo in increasing the time to the first occurrence of major adverse cardiovascular events (MACE) including coronary heart disease (CHD) death, ischemic stroke, myocardial infarction (MI), acute limb ischemia or major amputation, or urgent arterial revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following:

  1. Age ≥18 years with a history of a major atherosclerotic cardiovascular disease (ASCVD) event defined as at least 1 of the following: ≥30 days post MI (presumed Type 1 due to plaque rupture or erosion); ≥30 days post ischemic stroke (presumed due to atherosclerosis); or ≥30 days post successful peripheral (carotid or lower extremity) arterial revascularization (surgical or endovascular) or major (ankle or above) amputation due to atherosclerosis; or
  2. High risk for first major ASCVD event defined as at least 1 of the following: Age ≥50 years with evidence of coronary artery disease; Age ≥50 years with evidence of atherosclerotic cerebrovascular disease; Age ≥50 years with evidence of peripheral arterial disease; or Age ≥60 years with diabetes mellitus and at least one of the following: microvascular disease or urine albumin-creatinine ratio ≥30 mg/mmol within 6 months before Visit 1, daily insulin use, or diabetes for ≥10 years
* Has fasted lipid values (evaluated by the Central Laboratory) at Visit 1 (Screening) as follows:

  1. History of major ASCVD Event: LDL-C ≥70 mg/dL (1.81 mmol/L) OR non-HDL-C ≥100 mg/dL (2.59 mmol/L)
  2. High risk for first major ASCVD Event: LDL-C ≥90 mg/dL (2.33 mmol/L) OR non-HDL-C ≥120 mg/dL (3.11 mmol/L)
* Is treated with moderate- or high-intensity statin (± nonstatin lipid-lowering therapy [LLT]) at Visit 1
* Is on a stable dose of all background LLTs (including statin and nonstatin agents) for at least 30 days before Visit 1 (Screening) with no medication or dose changes planned during the participation in the study

Exclusion Criteria:

* Has a history of homozygous familial hypercholesterolemia (FH) based on genetic or clinical criteria, compound heterozygous FH, or double heterozygous FH
* Has New York Heart Association Class IV heart failure, last known Left Ventricular Ejection Fraction ≤25% by any imaging method, or had a Heart Failure hospitalization within 3 months before Visit 1 (Screening)
* Has recurrent ventricular tachycardia within 3 months prior to randomization
* Has a planned arterial revascularization procedure
* Is undergoing or previously underwent an LDL-C apheresis program within 3 months before Visit 1 (Screening) or plans to initiate an LDL-C apheresis program
* Was previously treated/is being treated with certain other cholesterol lowering medications, including protein convertase subtilisin/kexin type 9 (PCSK9) inhibitors without adequate washout.
* Has a fasting triglyceride value ≥400 mg/dL (≥4.52 mmol/L) at Visit 1 (Screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14550 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2029-11-29 (Estimated); Study Completion 2029-11-29 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Coronary Heart Disease (CHD) Death-Based Major Adverse Cardiovascular Events (MACE)-Plus | From date of randomization until the date of first occurrence of CHD death-based MACE-plus, assessed up to approximately 6 years
  Time to the first occurrence of CHD death-based MACE-plus, which is defined as any of the following: coronary heart disease death, myocardial infarction (MI), ischemic stroke (fatal and nonfatal), acute limb ischemia or major amputation, or urgent arterial revascularization (coronary, cerebrovascular, or peripheral).

SECONDARY OUTCOMES:
Time to First Occurrence of 3-point MACE | From date of randomization until the date of first occurrence of 3-point MACE, assessed up to approximately 6 years
  Time to the first occurrence of 3-point MACE (defined as cardiovascular death, MI, or ischemic stroke).
Time to First Occurrence of Cardiovascular (CV) Death-Based MACE Plus | From date of randomization until the date of first occurrence of CV death-based MACE plus, assessed up to approximately 6 years
  Time to the first occurrence of CV death-based MACE plus, defined as any of the following: cardiovascular death, MI, ischemic stroke, acute limb ischemia or major amputation, or urgent arterial revascularization (coronary, cerebrovascular, or peripheral).
Time to First Occurrence of CHD Death or MI | From date of randomization until the date of first occurrence of CHD death or MI, assessed up to approximately 6 years
  Time to the first occurrence of CHD death or MI.
Time to CV Death | From date of randomization until the date of CV death, assessed up to approximately 6 years
  Time to cardiovascular death.
Time to All-Cause Death | From date of randomization until the date of death, assessed up to approximately 6 years
  Time to all-cause death.
Time to CHD Death | From date of randomization until the date of CHD death, assessed up to approximately 6 years
  Time to CHD death.
Time to First Event of MI | From date of randomization until the date of MI, assessed up to approximately 6 years
  Time to the first occurrence of MI.
Time to First Event of Ischemic Stroke | From date of randomization until the date of first occurrence of ischemic stroke, assessed up to approximately 6 years
  Time to the first occurrence of ischemic stroke.
Time to First Event of Acute Limb Ischemia or Major Amputation | From date of randomization until the date of first occurrence of acute limb ischemia or major amputation, assessed up to approximately 6 years
  Time to the first occurrence of acute limb ischemia or major amputation.
Time to First Event of Urgent Arterial Revascularization | From date of randomization until the date of urgent arterial revascularization, assessed up to approximately 6 years
  Time to the first occurrence of urgent arterial revascularization (coronary, cerebrovascular, or peripheral).
Percent Change from Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline and Week 52
  The percent change from baseline in LDL-C.
Percent Change from Baseline in Apolipoprotein B | Baseline and Week 52
  The percent change from baseline in apolipoprotein B.
Percent Change from Baseline in Non-High-Density Lipoprotein Cholesterol (non-HDL-C) cholesterol | Baseline and Week 52
  The percent change from baseline in Non-HDL-C.
Percent Change from Baseline in Lipoprotein (a) | Baseline and Week 52
  The percent change from baseline in lipoprotein (a).
Number of Participants with an Adverse Event (AE) | Up to ~6 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with AE(s) in each arm will be reported.
Number of Participants Discontinuing from Study Therapy Due to AE | Up to ~6 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants discontinuing due to AE(s) in each arm will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (669):
- United States (132):
  - Advanced Cardiovascular - Alexander City ( Site 0156), Alexander City, Alabama
  - Central Research Associates ( Site 0118), Birmingham, Alabama
  - St. Vincent's Birmingham Hospital ( Site 0181), Birmingham, Alabama
  - Central Alabama Research ( Site 0109), Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC ( Site 0076), Daphne, Alabama
  - G&L Research ( Site 0042), Foley, Alabama
  - NextStage Clinical Research - Phoenix - (01) ( Site 0191), Glendale, Arizona
  - Synexus Clinical Research US, Inc.-Synexus Clinical Research US, Inc - Central Phoenix ( Site 0066), Phoenix, Arizona
  - Medical Investigations Inc. ( Site 0188), Little Rock, Arkansas
  - National Heart Institute-Research ( Site 0077), Beverly Hills, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI) ( Site 0130), La Jolla, California
  - Chemidox Clinical Trials ( Site 0145), Lancaster, California
  - Velocity Clinical Research, Westlake ( Site 0039), Los Angeles, California
  - Carbon Health - Pasadena ( Site 0149), Pasadena, California
  - Carbon Health - San Mateo - Hillsdale Mall ( Site 0151), San Mateo, California
  - America Clinical Trials-Research Dept ( Site 0104), Tarzana, California
  - Premiere Medical Center ( Site 0093), Toluca Lake, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center ( Site 0058), Torrance, California
  - University of Colorado Anschutz Medical Campus-University of Colorado Hospital Cardiac and Vascular ( Site 0146), Aurora, Colorado
  - South Denver Cardiology Associates ( Site 0167), Littleton, Colorado
  - Cardiology Associates of Fairfield County, P.C. ( Site 0159), Stamford, Connecticut
  - Chase Medical Research, LLC ( Site 0046), Waterbury, Connecticut
  - Emerson Clinical Research Institute ( Site 0143), Washington D.C., District of Columbia
  - Excel Medical Clinical Trials ( Site 0052), Boca Raton, Florida
  - Advanced Pharma Research ( Site 0040), Cutler Bay, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0083), Fort Myers, Florida
  - Westside Center for Clinical Research ( Site 0049), Jacksonville, Florida
  - University of Florida - Jacksonville ( Site 0166), Jacksonville, Florida
  - East Coast Institute for Research, LLC ( Site 0031), Jacksonville, Florida
  - Jacksonville Center for Clinical Research ( Site 0048), Jacksonville, Florida
  - East Coast Institute for Research ( Site 0034), Lake City, Florida
  - Columbus Clinical Services ( Site 0026), Miami, Florida
  - Miami Cardiac & Vascular Institute-Ambulatory Research ( Site 0059), Miami, Florida
  - Inpatient Research Clinic ( Site 0041), Miami Lakes, Florida
  - Eminat ( Site 0082), Miramar, Florida
  - Ocala Research Institute - Ocala - Southwest 20th Place ( Site 0079), Ocala, Florida
  - Progressive Medical Research ( Site 0045), Port Orange, Florida
  - St Johns Center for Clinical Research ( Site 0016), Saint Augustine, Florida
  - Clinical Site Partners LLC, dba CSP Orlando ( Site 0067), Winter Park, Florida
  - The Jones Center Clinical Research ( Site 0032), Macon, Georgia
  - North Georgia Clinical Research ( Site 0128), Woodstock, Georgia
  - Bingham Memorial Hospital ( Site 0195), Blackfoot, Idaho
  - Synexus Clinical Research US, Inc. ( Site 0084), Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood ( Site 0056), Chicago, Illinois
  - Great Lakes Clinical Trials - Gurnee ( Site 0134), Gurnee, Illinois
  - Alliance for Multispecialty Research, LLC ( Site 0173), Park Ridge, Illinois
  - Healthcare Research Network - Chicago ( Site 0051), Tinley Park, Illinois
  - Alliance for Multispecialty Research - Medisphere Medical Research Center ( Site 0080), Evansville, Indiana
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0154), Fort Wayne, Indiana
  - Franciscan Physician Network - Indiana Heart Physicians ( Site 0141), Indianapolis, Indiana
  - Reid Physician Associates ( Site 0174), Richmond, Indiana
  - University of Kansas Medical Center ( Site 0004), Kansas City, Kansas
  - Cotton O'Neil Clinical Research Center ( Site 0095), Topeka, Kansas
  - Alliance for Multispecialty Research, LLC ( Site 0116), Wichita, Kansas
  - Alliance for Multispecialty Research, LLC ( Site 0027), Lexington, Kentucky
  - L-MARC Research Center ( Site 0001), Louisville, Kentucky
  - Avant Research Associates ( Site 0103), Crowley, Louisiana
  - IMA Clinical Research- Monroe- North 18th Street ( Site 0111), Monroe, Louisiana
  - Northeast Cardiology Associates ( Site 0168), Bangor, Maine
  - Flourish Research - Bowie ( Site 0190), Bowie, Maryland
  - Centennial Medical Group ( Site 0179), Columbia, Maryland
  - Brigham and Women's Hospital-Cardiovascular Medicine ( Site 0147), Boston, Massachusetts
  - Boston Clinical Trials ( Site 0029), Boston, Massachusetts
  - Alliance for Multispecialty Research, LLC. ( Site 0171), Dearborn, Michigan
  - Healthy Heart Cardiology ( Site 0113), Grand Rapids, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division ( Site 0003), Troy, Michigan
  - Trinity Health-Michigan d/b/a Michigan Heart ( Site 0186), Ypsilanti, Michigan
  - Fairview Health Services ( Site 0024), Maplewood, Minnesota
  - Abbott Northwestern Hospital ( Site 0199), Minneapolis, Minnesota
  - University of Minnesota, Lillehei Clinical Research Unit ( Site 0193), Minneapolis, Minnesota
  - Velocity Clinical Research, Gulfport ( Site 0038), Gulfport, Mississippi
  - Cardiology Associates of North Mississippi ( Site 0169), Tupelo, Mississippi
  - Healthcare Research Network - St. Louis ( Site 0053), Hazelwood, Missouri
  - Alliance for Multispecialty Research, LLC ( Site 0071), Kansas City, Missouri
  - Skyline Medical Center/CCT Research ( Site 0148), Elkhorn, Nebraska
  - Velocity Clinical Research at The Pioneer Heart Institute, Lincoln ( Site 0078), Lincoln, Nebraska
  - CHI Health Clinic Heart Institute ( Site 0180), Lincoln, Nebraska
  - Excel Clinical Research, LLC ( Site 0123), Las Vegas, Nevada
  - Clinical Research of South Nevada ( Site 0135), Las Vegas, Nevada
  - Advanced Heart Care - Bridgewater Route 22 ( Site 0160), Bridgewater, New Jersey
  - Cardiovascular Associates of the Delaware Valley ( Site 0162), Washington Township, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center ( Site 0005), Albuquerque, New Mexico
  - Velocity Clinical Research, Binghamton ( Site 0063), Binghamton, New York
  - Central New York Clinical Research ( Site 0044), Manlius, New York
  - North Shore Diabetes & Endocrine Associates ( Site 0165), New Hyde Park, New York
  - Mid Hudson Medical Research ( Site 0087), New Windsor, New York
  - NYU Langone Health ( Site 0099), New York, New York
  - Rochester Clinical Research, Inc. ( Site 0098), Rochester, New York
  - Laurelton Heart Specialist PC ( Site 0092), Rosedale, New York
  - Duke University Health System (DUHS) ( Site 0153), Durham, North Carolina
  - Wake Forest Baptist Health-Cardiovascular Medicine ( Site 0142), Winston-Salem, North Carolina
  - Lillestol Research ( Site 0025), Fargo, North Dakota
  - Altru Health System ( Site 0197), Grand Forks, North Dakota
  - Velocity Clinical Research, Springdale ( Site 0112), Cincinnati, Ohio
  - Cleveland Clinic Main ( Site 0121), Cleveland, Ohio
  - The Ohio State Wexner Medical Center ( Site 0200), Columbus, Ohio
  - Remington-Davis, Inc. ( Site 0183), Columbus, Ohio
  - Premier Cardiovascular Institute ( Site 0136), Dayton, Ohio
  - Genesis Healthcare System-Pharmacy Research ( Site 0163), Zanesville, Ohio
  - South Oklahoma Heart Research ( Site 0164), Oklahoma City, Oklahoma
  - Capital Area Research, LLC ( Site 0139), Camp Hill, Pennsylvania
  - Guthrie Medical Group, P.C. ( Site 0176), Sayre, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley ( Site 0072), Yardley, Pennsylvania
  - Velocity Clinical Research, Anderson ( Site 0022), Anderson, South Carolina
  - Coastal Carolina Research Center ( Site 0006), North Charleston, South Carolina
  - Monument Health Clinical Research, a department of Monument -Monument Health Clinical Research, a d ( Site 0009), Rapid City, South Dakota
  - Holston Medical Group ( Site 0106), Bristol, Tennessee
  - Holston Medical Group ( Site 0047), Kingsport, Tennessee
  - Alliance for Multispecialty Research, LLC ( Site 0008), Knoxville, Tennessee
  - PharmaTex Research, LLC ( Site 0182), Amarillo, Texas
  - Texas Diabetes and Endocrinology, P.A. ( Site 0187), Austin, Texas
  - Southwest Family Medicine Associates ( Site 0189), Dallas, Texas
  - Prolato Clinical Research Center ( Site 0108), Houston, Texas
  - Permian Research Foundation ( Site 0157), Odessa, Texas
  - LinQ Research ( Site 0101), Pearland, Texas
  - Northeast Clinical Research of San Antonio ( Site 0011), San Antonio, Texas
  - Discovery Clinical Trials ( Site 0096), San Antonio, Texas
  - Sugar Lakes Family Practice, PA ( Site 0094), Sugar Land, Texas
  - LinQ Research - Tomball ( Site 0208), Tomball, Texas
  - Northwest Houston Heart Center-Northwest Houston Clinical Research, PLLC ( Site 0158), Tomball, Texas
  - NextStage Clinical Research - Waco ( Site 0196), Waco, Texas
  - Synexus Clinical Research US, Inc. ( Site 0086), Salt Lake City, Utah
  - Highland Clinical Research ( Site 0122), Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City ( Site 0019), West Jordan, Utah
  - Burke Internal Medicine and Research ( Site 0035), Burke, Virginia
  - Charlottesville Medical Research ( Site 0030), Charlottesville, Virginia
  - Virginia Heart ( Site 0097), Falls Church, Virginia
  - Carient Heart & Vascular - Manassas ( Site 0170), Manassas, Virginia
  - Manassas Clinical Research Center ( Site 0007), Manassas, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0043), Newport News, Virginia
  - Alliance for Multispecialty Research, LLC ( Site 0068), Norfolk, Virginia
  - Centricity Research Suffolk Family Medicine ( Site 0105), Suffolk, Virginia
- Argentina (21):
  - CEDIC ( Site 0612), CABA, Buenos Aires
  - CEMEDIC ( Site 0609), CABA, Buenos Aires
  - Framingham Centro Médico ( Site 0625), La Plata, Buenos Aires
  - CIMeL ( Site 0613), Lanús, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0605), Mar del Plata, Buenos Aires
  - DIM Clínica Privada ( Site 0627), Ramos Mejía, Buenos Aires
  - Go Centro Medico San Nicolás ( Site 0621), San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate ( Site 0600), Zárate, Buenos Aires
  - CIPREC-CIPREC Sede Arenales ( Site 0624), Buenos Aires, Buenos Aires F.D.
  - Fundación favaloro para la Docencia e Investigación Médica ( Site 0606), Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada ( Site 0604), Buenos Aires, Buenos Aires F.D.
  - Fundación Respirar ( Site 0610), Buenos Aires, Buenos Aires F.D.
  - Instituto Médico DAMIC ( Site 0603), Córdoba, Córdoba Province
  - Instituto de Investigaciones Clinicas Rosario ( Site 0602), Rosario, Santa Fe Province
  - Fundacion Estudios Clinicos ( Site 0619), Rosario, Santa Fe Province
  - Laboratorio de Hemostasia y Trombosis ( Site 0623), Rosario, Santa Fe Province
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares ( Site 0615), Santa Fe, Santa Fe Province
  - Sanatorio Finochietto ( Site 0626), Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME) ( Site 0620), CABA
  - Instituto de Cardiología "Juana F. Cabral"-Cardiología ( Site 0608), Corrientes
  - Centro de Investigaciones Clinicas del Litoral ( Site 0607), Santa Fe
- Australia (7):
  - Paratus Clinical Research Canberra ( Site 2804), Bruce, Australian Capital Territory
  - Paratus Clinical Research Western Sydney ( Site 2805), Blacktown, New South Wales
  - Royal Prince Alfred Hospital ( Site 2808), Camperdown, New South Wales
  - Paratus Clinical Research Central Coast ( Site 2806), Kanwal, New South Wales
  - The Prince Charles Hospital ( Site 2810), Brisbane, Queensland
  - Victorian Heart Hospital-Monash Cardiovascular Research Centre (MCRC) ( Site 2803), Clayton, Victoria
  - Baker IDI Heart & Diabetes Institute ( Site 2809), Hoppers Crossing, Victoria
- Brazil (18):
  - Centro de Pesquisas em Diabetes e Doenças Endócrino-Metabólicas ( Site 0728), Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Brasil ( Site 0719), Brasília, Federal District
  - Universidade Federal de Goias ( Site 0717), Goiânia, Goiás
  - Hospital Angelina Caron ( Site 0702), Campina Grande do Sul, Paraná
  - Hospital do Rocio ( Site 0721), Campo Largo, Paraná
  - Hospital Universitário ( Site 0723), Canoas, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul ( Site 0704), Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus ( Site 0716), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição-FZ PESQUISA E SERVIÇOS EM CARDIOLOGIA CLÍNICA LTDA ( Site 0712), Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clinica do Coracao ( Site 0713), Aracaju, Sergipe
  - Hospital Universitário São Francisco de Assis - Bragança Paulista ( Site 0725), Bragança Paulista, São Paulo
  - Instituto de Pesquisa clinica de Campinas ( Site 0706), Campinas, São Paulo
  - Hospital e Maternidade Christóvão da Gama (HMCG) ( Site 0724), Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0707), São José do Rio Preto, São Paulo
  - Instituto Dante Pazzanese de Cardiology-Fundação Adib Jatene ( Site 0708), São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica ( Site 0710), São Paulo, São Paulo
  - Integral Pesquisa e Ensino ( Site 0709), Votuporanga, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica ( Site 0715), Rio de Janeiro
- Canada (10):
  - OCT Research ULC ( Site 0512), Kelowna, British Columbia
  - Cambridge Cardiac Care Centre ( Site 0508), Cambridge, Ontario
  - North York Diagnostic and Cardiac Centre ( Site 0514), North York, Ontario
  - Oakville Cardiovascular Research LP ( Site 0507), Oakville, Ontario
  - Corcare ( Site 0511), Toronto, Ontario
  - Ecogene-21 ( Site 0510), Chicoutimi, Quebec
  - Institut de Cardiologie de Montreal ( Site 0506), Montreal, Quebec
  - IUCPQ ( Site 0515), Québec, Quebec
  - Centre intégré de santé et de services sociaux de Lanaudière - Hopital Pierre-Le Gardeur. ( Site 0509), Terrebonne, Quebec
  - Diex Recherche Trois-Rivieres ( Site 0505), Trois-Rivières, Quebec
- Chile (15):
  - Clinical Research Chile SpA ( Site 0804), Valdivia, Los Ríos Region
  - Centro de Investigación del Maule ( Site 0816), Talca, Maule Region
  - Espacio Eme ( Site 0806), Ñuñoa, Region M. de Santiago
  - Servicios Medicos Godoy ( Site 0810), Providencia, Region M. de Santiago
  - Enroll SpA ( Site 0803), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 0815), Santiago, Region M. de Santiago
  - CECIM ( Site 0811), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinicadela Universidad Catolica ( Site 0812), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile ( Site 0800), Santiago, Region M. de Santiago
  - Clínica Ensenada ( Site 0801), Santiago, Region M. de Santiago
  - Centro de Investigación Clinica Del Sur ( Site 0821), Temuco, Región de la Araucanía
  - Centro De Estudios Cardiologicos Y De Medicina Interna ( Site 0805), Temuco, Región de la Araucanía
  - Centro Respiratorio Integral - CENRESIN. ( Site 0820), Quillota, Región de Valparaíso
  - ONCOCENTRO APYS ( Site 0808), Viña del Mar, Región de Valparaíso
  - Biocenter ( Site 0819), Concepción, Región del Biobío
- China (58):
  - Second Affiliated hospital of Anhui Medical University-Cardiology ( Site 3458), Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University-Cardiovascular ( Site 3400), Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital ( Site 3423), Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University ( Site 3424), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 3441), Chongqing, Chongqing Municipality
  - The Eighth Affiliated Hospital of Southern Medical University ( Site 3427), Foshan, Guangdong
  - Guangdong Provincial People's Hospital-Cardiology ( Site 3402), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University ( Site 3415), Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital ( Site 3467), Huizhou, Guangdong
  - Jiangmen Center Hospital ( Site 3492), Jiangmen, Guangdong
  - The University of Hong Kong-Shenzhen Hospital-Cardiovascular department ( Site 3414), Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University ( Site 3486), Guiyang, Guizhou
  - Hainan General Hospital ( Site 3409), Haikou, Hainan
  - Daqing People's Hospital-Cardiology ( Site 3470), Daqing, Heilongjiang
  - The first affiliated Hospital of Harbin Medical University-Cardiology ( Site 3406), Harbin, Heilongjiang
  - The Fourth Hospital of Harbin Medical University-Endocrinology department ( Site 3452), Harbin, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical University ( Site 3465), Qiqihar, Heilongjiang
  - Nanyang First People's Hospital ( Site 3469), Nanyang, Henan
  - Pu'ai Hospital of Wuhan City ( Site 3451), Wuhan, Hubei
  - Renmin Hospital of Wuhan University ( Site 3464), Wuhan, Hubei
  - Changsha Central Hospital-Cardiovascular ( Site 3404), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University-Cardiology ( Site 3412), Changsha, Hunan
  - The Third Hospital of Changsha-Cardiovascular department ( Site 3434), Changsha, Hunan
  - The First People's Hospital of Yueyang-Cardiovascular department ( Site 3448), Yueyang, Hunan
  - Baotou Central Hospital-Cardiology ( Site 3436), Baotou, Inner Mongolia
  - Chifeng Hospital-Department of Cardiology ( Site 3433), Chifeng, Inner Mongolia
  - Inner Mongolia People's Hospital ( Site 3439), Hohhot, Inner Mongolia
  - Changzhou Second People's Hospital-Cardiology ( Site 3459), Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Cardiology ( Site 3480), Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 3403), Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital ( Site 3405), Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University-Cardiology Department ( Site 3481), Zhenjiang, Jiangsu
  - The Third Hospital of Nanchang - Fuhe-cardiology ( Site 3496), Nanchang, Jiangxi
  - The Third Hospital of Nanchang ( Site 3454), Nanchang, Jiangxi
  - Pingxiang People's Hospital-Cardiology ( Site 3473), Pingxiang, Jiangxi
  - Jilin Province People's Hospital-Department of Cardiology ( Site 3442), Changchun, Jilin
  - Siping Central People's Hospital-Cardiovascular Department ( Site 3408), Siping, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University ( Site 3476), Jinzhou, Liaoning
  - The People's Hospital of Liaoning Province-Cardiology ( Site 3453), Shenyang, Liaoning
  - General Hospital of Ningxia Medical University ( Site 3478), Yinchuan, Ningxia
  - Shanxi Cardiovascular Hospital ( Site 3462), Taiyuan, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 3420), Xi'an, Shaanxi
  - Shaanxi provincial people's hospital ( Site 3421), Xi'an, Shaanxi
  - Xianyang Hospital of Yan'an University ( Site 3435), Xianyang, Shaanxi
  - Linyi People's Hospital ( Site 3468), Linyi, Shandong
  - Zibo Municipal Hospital ( Site 3474), Zibo, Shandong
  - Shanghai Tongji Hospital ( Site 3431), Shanghai, Shanghai Municipality
  - Shanghai General Hospital ( Site 3479), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 3485), Shanghai, Shanghai Municipality
  - The Third People's Hospital of Chengdu (CDTPH) ( Site 3430), Chengdu, Sichuan
  - Chengdu Second Municipal People's Hospital ( Site 3419), Chengdu, Sichuan
  - The Second People's Hospital of Neijiang ( Site 3482), Neijiang, Sichuan
  - Suining Central Hospital ( Site 3487), Suining, Sichuan
  - Tianjin People' s Hospital-Cardiology ( Site 3425), Tianjin, Tianjin Municipality
  - Tianjin Fourth Centre Hospital-Department of Cardiology ( Site 3456), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 3417), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province-Cardiovascular Department ( Site 3472), Linhai, Zhejiang
  - Lishui Central Hospital ( Site 3455), Lishui, Zhejiang
- Colombia (18):
  - Fundación Centro de Investigación Clínica CIC ( Site 0906), Medellín, Antioquia
  - Salud SURA Industriales ( Site 0917), Medellín, Antioquia
  - Rodrigo Botero S.A.S ( Site 0901), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 0903), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 0902), Barranquilla, Atlántico
  - IPS Centro Científico Asistencial S.A.S ( Site 0900), Barranquilla, Atlántico
  - IPS Médicos Internistas de Caldas ( Site 0905), Manizales, Caldas Department
  - Instituto Cardiovascular del Cesar S.A ( Site 0919), Valledupar, Cesar Department
  - Sociedad de Cirugía de Bogotá - Hospital de San Jose ( Site 0920), Bogota, Cundinamarca
  - Fundacion Santa Fe de Bogota ( Site 0916), Bogotá, Cundinamarca
  - Solano & Terront Servicios Medicos - UNIENDO ( Site 0915), Bogotá, Cundinamarca
  - Salud SURA Calle 100 ( Site 0918), Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S ( Site 0913), Zipaquirá, Cundinamarca
  - IMAT S.A.S ( Site 0907), Montería, Departamento de Córdoba
  - Fundación Cardiovascular de Colombia ( Site 0911), Piedecuesta, Santander Department
  - Mediservis del Tolima IPS S.A.S ( Site 0914), Ibagué, Tolima Department
  - Fundación Valle del Lili ( Site 0904), Cali, Valle del Cauca Department
  - Centro de Investigaciones Clinicas SAS ( Site 0912), Cali, Valle del Cauca Department
- Denmark (11):
  - Herlev and Gentofte Hospital-Department of Cardiology ( Site 1210), Copenhagen, Capital Region
  - Sanos Clinic-Sanos Clinic ( Site 1204), Herlev, Capital Region
  - Aarhus Universitetshospital, Skejby ( Site 1201), Aarhus, Central Jutland
  - Regionshospitalet Gødstrup ( Site 1207), Herning, Central Jutland
  - Sanos Clinic - Nordjylland ( Site 1203), Gandrup, North Denmark
  - Sygehus Vendsyssel Hjoerring ( Site 1209), Hjørring, North Denmark
  - Roskilde Sygehus ( Site 1212), Roskilde, Region Sjælland
  - Slagelse Sygehus-Ambulatorium for Hjertesygdomme ( Site 1205), Slagelse, Region Sjælland
  - Sydvestjysk Sygehus Esbjerg ( Site 1206), Esbjerg, Region Syddanmark
  - Svendborg Hospital Odense Universitets hospital-Kardiologisk Forskningsenhed ( Site 1200), Svendborg, Region Syddanmark
  - Sanos Clinic - Syddanmark ( Site 1202), Vejle, Region Syddanmark
- France (15):
  - Centre Hospitalier Universitaire de Grenoble-Cardiology ( Site 1421), Grenoble, Auvergne-Rhône-Alpes
  - CHRU Troussau-CARDIOLOGY ( Site 1402), Chambray-lès-Tours, Centre-Val de Loire
  - CENTRE HOSPITALIER REGIONAL D'ORLEANS-Service de Cardiologie ( Site 1416), Orléans, Centre-Val de Loire
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 1409), Dijon, Cote-d Or
  - Centre Hospitalier Louis Pasteur ( Site 1405), Le Coudray, Eure-et-Loir
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Universitaire Carémeau ( Site 1401), Nîmes, Gard
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren ( Site 1413), Limoges, Haute-Vienne
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou ( Site 1404), Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire de Reims - Hôpital Robert Debré ( Site 1418), Reims, Marne
  - Polyclinique Vauban ( Site 1406), Valenciennes, Nord
  - Pitie Salpetriere University Hospital ( Site 1414), Paris, Orne
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord ( Site 1400), Saint Priest En Jarez, Pays de la Loire Region
  - Centre Hospitalier de Pau ( Site 1408), Pau, Pyrenees-Atlantiques
  - Clinique du Pont de Chaume ( Site 1407), Montauban, Tarn-et-Garonne
  - Centre Hospitalier Universitaire de Poitiers ( Site 1417), Poitiers, Vienne
- Germany (30):
  - Klinikum am Plattenwald ( Site 1590), Bad Friedrichshall, Baden-Wurttemberg
  - Siteworks GmbH - Heidelberg ( Site 1546), Heidelberg, Baden-Wurttemberg
  - ze:ro ARZTPRAXEN-Ze:ro Praxen ( Site 1583), Mannheim, Baden-Wurttemberg
  - Kardiologische Gemeinschaftspraxis ( Site 1564), Nuremberg, Bavaria
  - Gemeinschaftspraxis Dr. med. Josef und Wilma Großkopf ( Site 1547), Wallerfing, Bavaria
  - Kerckhoff-Klinik ( Site 1599), Bad Nauheim, Hesse
  - Synexus Clinical Research GmbH Synexus Frankfurt Clinical Research Centre ( Site 1592), Frankfurt am Main, Hesse
  - ClinPhenomics CVC GmbH ( Site 1593), Frankfurt am Main, Hesse
  - Siteworks GmbH ( Site 1552), Hanover, Lower Saxony
  - Studienzentrum Brinkum - Torsten Drescher & Dr. Lars Pohlmeier ( Site 1557), Stuhr, Lower Saxony
  - Klinikum Bielefeld Mitte ( Site 1561), Bielefeld, North Rhine-Westphalia
  - Zentrum fur klinische Forschung - Köln ( Site 1573), Cologne, North Rhine-Westphalia
  - St.-Johannes-Hospital Dortmund-Clinic of Internal medicine I ( Site 1567), Dortmund, North Rhine-Westphalia
  - Die Bocholder Hausärzte ( Site 1587), Essen, North Rhine-Westphalia
  - Klinisches Forschungszentrum Dr. Hagemann am Hausarztzentrum am Germaniaplatz ( Site 1554), Essen, North Rhine-Westphalia
  - Unterfrintroper Hausarztzentrum Klinische Forschung ( Site 1550), Essen, North Rhine-Westphalia
  - Forschungszentrum Ruhr ( Site 1586), Witten, North Rhine-Westphalia
  - Kardiopraxis Schirmer Kaiserslautern ( Site 1576), Kaiserslautern, Rhineland-Palatinate
  - Siteworks GmbH - Völklingen ( Site 1553), Völklingen, Saarland
  - Zentrum fuer klinische Pruefungen in der Facharztzentrum Dresden Neustadt GbR ( Site 1597), Dresden, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden-Universitätsstudienzentrum für Stoffwechselerkranku ( Site 1549), Dresden, Saxony
  - Synexus Leipzig Clinical Research Centre ( Site 1591), Leipzig, Saxony
  - Hausarzt- und Diabetologische Schwerpunktpraxis Hohenmölsen - Weiβenfels ( Site 1574), Hohenmölsen, Saxony-Anhalt
  - Praxis Rankestrasse ( Site 1548), Berlin
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin ( Site 1568), Berlin
  - DRK Kliniken Berlin - Köpenick ( Site 1580), Berlin
  - Synexus Berlin Clinical Research Centre ( Site 1585), Berlin
  - Jüdisches Krankenhaus Berlin ( Site 1595), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 1556), Hamburg
  - Cardiologicum Hamburg ( Site 1596), Hamburg
- Hong Kong (5):
  - Queen Mary Hospital-Medicine - Cardiology ( Site 3303), Hksar
  - Queen Mary Hospital-Medical ( Site 3300), Pok Fu Lam
  - Prince of Wales Hospital ( Site 3301), Shatin
  - Prince of Wales Hospital ( Site 3304), Shatin
  - Our Lady of Maryknoll Hospital-Department of Medicine and Geriatrics ( Site 3305), Wong Tai Sin
- Hungary (17):
  - Private Practice - Dr. Lakatos Ferenc ( Site 1618), Békéscsaba, Bekes County
  - Lausmed Egészségügyi Szolgáltató ( Site 1621), Baja, Bács-Kiskun county
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Belgyógyászati Klinika ( Site 1617), Szeged, Csongrád megye
  - Fejér Megyei Szent György Egyetemi Oktató Kórház-2nd Department of Internal Medicine ( Site 1611), Székesfehérvár, Fejér
  - Belinus Orvosi és Számitástechnikai Bt ( Site 1608), Debrecen, Hajdú-Bihar
  - CoroMed ( Site 1612), Pécs, Pecs
  - Óbudai Egészségügyi Centrum - Kaposvár Site ( Site 1625), Kaposvár, Somogy County
  - Borbánya Praxis-Private practice ( Site 1606), Nyíregyháza, Borbánya, Szabolcs-Szatmár-Bereg
  - DRC Gyógyszervizsgáló Központ ( Site 1609), Balatonfüred, Veszprém megye
  - Zuglói Egészségügyi Szolgálat ( Site 1613), Budapest, Zala County
  - Óbudai Egészségügyi Centrum ( Site 1622), Budapest
  - Gottsegen György Országos Kardiovaszkuláris Intézet ( Site 1605), Budapest
  - Semmelweis Egyetem-Városmajori Szív- és Érgyógyászati Klinika ( Site 1601), Budapest
  - Medoc Egészégközpont - Lehel ( Site 1615), Budapest
  - Cardiogeneral Egészségügyi Kft. ( Site 1610), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Anyagcsere Tanszék) ( Site 1607), Debrecen
  - Óbudai Egészségügyi Centrum - Zalaegerszeg ( Site 1624), Zalaegerszeg
- Israel (18):
  - Barzilai Medical Center ( Site 1713), Ashkelon
  - Soroka Medical Center ( Site 1715), Beersheba
  - Hillel Yaffe Medical Center ( Site 1705), Hadera
  - Linn Medical Center ( Site 1711), Haifa
  - Rambam Health Care Campus ( Site 1702), Haifa
  - Rambam Health Care Campus ( Site 1718), Haifa
  - Institute of Diabetes, Technology and Research - Clalit Health ( Site 1701), Herzliya
  - Clalit health Services - Holon Medical Center ( Site 1721), Holon
  - Shaare Zedek Medical Center ( Site 1710), Jerusalem
  - Hadassah Medical Center ( Site 1706), Jerusalem
  - Hadassah Medical Center ( Site 1709), Jerusalem
  - Clalit Health Services - Majd Al-Krum Clinic ( Site 1722), Majd el Kurūm
  - Galilee Medical Center ( Site 1723), Nahariya
  - Rabin Medical Center ( Site 1720), Petah Tikva
  - Rabin Medical Center ( Site 1703), Petah Tikva
  - Sheba Medical Center ( Site 1708), Ramat Gan
  - Kaplan Medical Center ( Site 1724), Rehovot
  - Clalit Health Services - Sakhnin Community Clinic-Research Unit ( Site 1700), Sakhnin
- Italy (17):
  - Azienda Ospedaliero Universitaria di Ferrara ( Site 1816), Cona, Ferrara
  - Fondazione Policlinico Universitario Campus Bio-Medico ( Site 1818), Rome, Lazio
  - Fondazione Policlinico Tor Vergata ( Site 1809), Rome, Lazio
  - AOU Policlinico Umberto I-Dipartimento di Scienze Cliniche, Internistiche, Anestesiologiche e Cardi ( Site 1808), Rome, Lazio
  - Policlinico Gemellli - UOC di cardiologia ( Site 1821), Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII-Cardiologia 1 ( Site 1817), Bergamo, Lombardy
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia ( Site 1820), Brescia, Lombardy
  - Centro Cardiologico Monzino ( Site 1804), Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda-Unità Ricerche Cliniche della Cardiologia 4 ( Site 1811), Milan, Milano
  - Policlinico di Monza centro diabetologia e malattie metaboliche ( Site 1806), Monza, Monza E Brianza
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino ( Site 1801), Turin, Piedmont
  - A.O.U. Policlinico Paolo Giaccone ( Site 1815), Palermo, Sicily
  - ASST DI LECCO ( Site 1814), Lecco
  - University of Naples Federico II ( Site 1805), Napoli
  - Azienda Ospedaliero Universitaria di Parma ( Site 1813), Parma
  - Fondazione IRCCS Policlinico San Matteo-Cardiology ( Site 1802), Pavia
  - Ospedale Mauriziano ( Site 1812), Torino
- Japan (38):
  - Nagoya Kyoritsu Hospital ( Site 3531), Nagoya, Aichi-ken
  - Chubu Rosai Hospital ( Site 3507), Nagoya, Aichi-ken
  - Toyota Kosei Hospital ( Site 3519), Toyota, Aichi-ken
  - Toyota Memorial Hospital ( Site 3539), Toyota, Aichi-ken
  - Seikeikai Medical Corporation New Tokyo Heart Clinic ( Site 3537), Matsudo, Chiba
  - Nakamura Cardiovascular Clinic ( Site 3529), Itoshima, Fukuoka
  - Fukuoka Tokushukai Hospital ( Site 3511), Kasuga, Fukuoka
  - Kokura Memorial Hospital ( Site 3521), Kitakyushu, Fukuoka
  - Go Neurosurgical Clinic ( Site 3534), Nakagawa, Fukuoka
  - Matsuda Cardiovascular Clinic ( Site 3526), Sapporo, Hokkaido
  - Hyogo Prefectural Harima-Himeji General Medical Center ( Site 3514), Himeji, Hyōgo
  - Tsukuba Medical Center Hospital ( Site 3540), Tsukuba, Ibaraki
  - TAKAMATSU Red Cross Hospital ( Site 3506), Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital ( Site 3538), Takamatsu, Kagawa-ken
  - Fujisawa City Hospital ( Site 3522), Fujisawa, Kanagawa
  - Tokai University Hospital ( Site 3500), Isehara, Kanagawa
  - Shonan Kamakura General Hospital ( Site 3516), Kamakura, Kanagawa
  - Kyoto Okamoto Memorial Hospital ( Site 3524), Kuse-gun Kumiyama-cho, Kyoto
  - Uji-Tokushukai Medical Center ( Site 3509), Uji, Kyoto
  - National Hospital Organization Nagasaki Medical Center ( Site 3505), Ōmura, Nagasaki
  - Saga-Ken Medical Centre Koseikan ( Site 3543), Saga, Saga-ken
  - Hanyu General Hospital ( Site 3504), Hanyū, Saitama
  - Tokyonishi Tokushukai Hospital ( Site 3530), Akishima, Tokyo
  - Minamino Cardiovascular Hospital ( Site 3546), Hachiōji, Tokyo
  - Affiliated Central Clinic of Higashiyamato Hospital ( Site 3533), Higashiyamato, Tokyo
  - Saiseikai Fukuoka General Hospital ( Site 3536), Fukuoka
  - Fukuoka University Hospital ( Site 3502), Fukuoka
  - Japanese Red Cross Fukuoka Hospital ( Site 3528), Fukuoka
  - Kumamoto University Hospital ( Site 3501), Kumamoto
  - Saiseikai Kumamoto Hospital ( Site 3515), Kumamoto
  - Kyoto City Hospital ( Site 3542), Kyoto
  - Nagasaki Harbor Medical Center ( Site 3527), Nagasaki
  - Okayama City General Medical Center Okayama City Hospital ( Site 3508), Okayama
  - National Hospital Organization Okayama Medical Center ( Site 3512), Okayama
  - National Hospital Organization Osaka National Hospital ( Site 3503), Osaka
  - Sanai Hospital - Saitama ( Site 3532), Saitama
  - Saitama City Hospital ( Site 3535), Saitama
  - Machida Municipal Hospital ( Site 3545), Tokyo
- Mexico (30):
  - Centro de Investigacion Cardiovascular y Metabólica ( Site 1027), Tijuana, Estado de Baja California
  - Morales Vargas Centro de Investigacion ( Site 1029), León, Guanajuato
  - Grupo Ollin Care ( Site 1023), Pachuca, Hidalgo
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad-Endocrinology ( Site 1007), Guadalajara, Jalisco
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occident-Unidad de Investigación Clínica Cardio ( Site 1015), Guadalajara, Jalisco
  - Cardiocent de Guadalajara S.C.-cardiocent de guadalajara SC ( Site 1001), Guadalajara, Jalisco
  - Centro de Investigación Médico Biológica y Terapia Avanzada ( Site 1021), Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente, S.C.-Departamento de Centro de Investigacion Medica d ( Site 1022), Zapopan, Jalisco
  - HOSPITAL GENERAL DE MEXICO DR. EDUARDO LICEAGA-Farmacologia Clinica ( Site 1033), Mexico City, Mexico City
  - Centro de Imagen y Tecnología en Intervención Cardiovascular-Research ( Site 1041), Mexico City, Mexico City
  - Bio Investigación AMARC, S.C. ( Site 1013), Mexico City, Mexico City
  - Clínica Integral del Paciente Diabético y Obeso ( Site 1016), Mexico City, Mexico City
  - Medica Sur-Clinica de Enfermedades Digestivas y Obesidad ( Site 1024), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 1012), Mexico City, Mexico City
  - CHRISTUS Centro de Excelencia en Investigación (Norte) ( Site 1032), General Escobedo, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Endocrinologia ( Site 1025), Monterrey, Nuevo León
  - Unidad biomedica avanzada monterrey-Clinical Trials ( Site 1000), Monterrey, Nuevo León
  - Centro de investigación y control metabólico ( Site 1003), Monterrey, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C. ( Site 1006), Ciudad Madero, Tamaulipas
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan ( Site 1017), Mérida, Yucatán
  - Centro de Atención e Investigación Clínica ( Site 1010), Aguascalientes
  - Centro de Investigación Cardiometabólica de Aguascalientes ( Site 1034), Aguascalientes
  - Fundación Cardiovascular de Aguascalientes A.C. ( Site 1020), Aguascalientes
  - ICARO Investigaciones en Medicina ( Site 1005), Chihuahua City
  - Centro de Investigación y Gastroenterología ( Site 1002), Cuauhtémoc
  - Instituto Nacional de Cardiologia Ignacio Chavez-Endocrinology ( Site 1018), México
  - Oaxaca Site Management Organization S.C. ( Site 1004), Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca ( Site 1011), Oaxaca City
  - Instituto Veracruzano en Investigación Clínica S.C. ( Site 1035), Veracruz
  - Arké SMO S.A de C.V ( Site 1026), Veracruz
- Netherlands (35):
  - Treant, locatie Scheper Ziekenhuis ( Site 1918), Emmen, Drenthe
  - Treant, locatie Ziekenhuis Bethesda-Bethesda Diabetes Research Center ( Site 1930), Hoogeveen, Drenthe
  - Gelre Ziekenhuis ( Site 1907), Apeldoorn, Gelderland
  - Slingeland Ziekenhuis ( Site 1941), Doetinchem, Gelderland
  - Ziekenhuis Gelderse Vallei ( Site 1939), Ede, Gelderland
  - Ziekenhuis St. Jansdal ( Site 1917), Harderwijk, Gelderland
  - Radboudumc-Cardiology ( Site 1925), Nijmegen, Gelderland
  - Ziekenhuis Rivierenland-Remati ( Site 1916), Tiel, Gelderland
  - Gelre Ziekenhuizen ( Site 1908), Zutphen, Gelderland
  - VieCuri Medisch Centrum, locatie Venlo-Cardiology ( Site 1923), Venlo, Limburg
  - Amphia Ziekenhuis, locatie Breda Molengracht-Research cardiology ( Site 1903), Breda, North Brabant
  - Catharina Ziekenhuis ( Site 1934), Eindhoven, North Brabant
  - Elkerliek Ziekenhuis ( Site 1938), Helmond, North Brabant
  - Bravis Ziekenhuis, locatie Roosendaal ( Site 1905), Roosendaal, North Brabant
  - Noordwest Ziekenhuisgroep-Research Cardiology ( Site 1914), Alkmaar, North Holland
  - Ziekenhuis Amstelland-Cardiologie ( Site 1920), Amstelveen, North Holland
  - Onze Lieve Vrouwe Gasthuis ( Site 1922), Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC-Vascular Medicine Clin Trial Unit ( Site 1926), Amsterdam, North Holland
  - Tergooiziekenhuizen, locatie Hilversum ( Site 1929), Hilversum, North Holland
  - Dijklander Ziekenhuis ( Site 1936), Hoorn, North Holland
  - Zaans Medisch Centrum ( Site 1942), Zaandam, North Holland
  - Ziekenhuisgroep Twente, locatie Almelo-Cardioresearch ZGT ( Site 1919), Almelo, Overijssel
  - Medische Centrum Leeuwarden ( Site 1935), Leeuwarden, Provincie Friesland
  - Antonius Ziekenhuis, locatie D&A Research and Genetics ( Site 1928), Sneek, Provincie Friesland
  - Reinier de Graaf Ziekenhuis, locatie Delft-Research Department Cardiology ( Site 1915), Delft, South Holland
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk ( Site 1901), Dordrecht, South Holland
  - Groene Hart Ziekenhuis-Research Cardiologie ( Site 1932), Gouda, South Holland
  - Leids Universitair Medisch Centrum ( Site 1924), Leiden, South Holland
  - Alrijne Ziekenhuis, locatie Leiderdorp ( Site 1902), Leiderdorp, South Holland
  - Erasmus Medisch Centrum, Centrumlocatie ( Site 1943), Rotterdam, South Holland
  - Ikazia Ziekenhuis ( Site 1911), Rotterdam, South Holland
  - Haga Ziekenhuis locatie Leyweg ( Site 1909), The Hague, South Holland
  - Meander Medisch Centrum ( Site 1933), Amersfoort, Utrecht
  - Admiraal de Ruyter Ziekenhuis, locatie Goes ( Site 1900), Goes, Zeeland
  - Martini Ziekenhuis ( Site 1940), Groningen
- New Zealand (16):
  - Pacific Clinical Research Network - Rotorua ( Site 2902), Rotorua, Bay of Plenty
  - Momentum Clinical Research - Tauranga ( Site 2907), Tauranga, Bay of Plenty
  - New Zealand Clinical Research (Christchurch) ( Site 2901), Christchurch, Canterbury
  - Pacific Clinical Research Network - Forte ( Site 2903), Christchurch, Canterbury
  - Momentum Clinical Research Hawke's Bay ( Site 2913), Hastings, Hawkes Bay
  - Momentum Clinical Research - Palmerston North ( Site 2909), Palmerston North, Manawatu-Wanganui
  - Momentum Clinical Research Dunedin ( Site 2910), Dunedin, Otago
  - Lakeland Clinical Trials Waikato ( Site 2906), Nawton, Waikato Region
  - Lakeland Clinical Trials Wellington ( Site 2904), Ebdentown, Wellington Region
  - Momentum Clinical Research Lower Hutt ( Site 2914), Lower Hutt, Wellington Region
  - Waitemata District Health Board ( Site 2915), Auckland
  - New Zealand Clinical Research (Auckland) ( Site 2900), Auckland
  - Waitemata Clinical Research Ltd ( Site 2916), Auckland
  - Auckland City Hospital ( Site 2911), Auckland
  - Pacific Clinical Research Network - Tasman ( Site 2905), Nelson
  - Momentum Clinical Research Kapiti ( Site 2912), Wellington
- Norway (9):
  - Akershus Universitetssykehus-Hjertemedisinsk Avdeling ( Site 2028), Lorenskog, Akershus
  - Haukeland Universitetssjukehus ( Site 2023), Bergen, Hordaland
  - Ålesund sjukehus ( Site 2029), Ålesund, Møre og Romsdal
  - Nordlandssykehuset ( Site 2021), Bodø, Nordland
  - Sykehuset Innlandet HF Lillehammer-Medisinsk avdeling ( Site 2030), Lillehammer, Oppland
  - Oslo Universitetssykehus Aker-Lipidklinikken ( Site 2020), Oslo
  - Colosseumsklinikken AS ( Site 2024), Oslo
  - Oslo Universitetssykehus Rikshospitalet-Kardiologisk avdeling ( Site 2025), Oslo
  - Oslo Universitetssykehus Ullevål ( Site 2031), Oslo
- Peru (17):
  - Hogar Clínica San Juan de Dios ( Site 1115), Arequipa, Ariqipa
  - Centro de investigacion Clínica Trujillo-Medical specialties ( Site 1104), Trujillo, La Libertad
  - Clínica San Antonio ( Site 1118), Trujillo, La Libertad
  - Policlínico Especializado en Neurología ( Site 1112), La Perla-Callao, Lima
  - ASOCIACION CIVIL POR LA SALUD ( Site 1107), Miraflores, Muni Metro de Lima
  - Hospital Alberto Sabogal Sologuren ( Site 1109), Bellavista, Qallaw
  - Unidad de Investigacon de la Clinica Internacional ( Site 1116), Lima
  - Clínica Internacional - Sede San Borja ( Site 1111), Lima
  - Clínica Vesalio-Cardiology ( Site 1101), Lima
  - Clínica Javier Prado ( Site 1100), Lima
  - Hospital Militar Geriátrico ( Site 1114), Lima
  - CLINICA DELGADO ( Site 1117), Lima
  - Clínica El Golf-Cardiologia ( Site 1103), Lima
  - Clínica Providencia ( Site 1102), Lima
  - Hospital Cayetano Heredia-Servicio de cardiologia ( Site 1113), Lima
  - Centro de Investigación Clínica Belén ( Site 1108), Piura
  - Instituto Médico Soy Diabetico ( Site 1106), Piura
- Poland (32):
  - Solumed Centrum Medyczne ( Site 2123), Poznan, Greater Poland Voivodeship
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością MEDIC-R Sp.k ( Site 2150), Poznan, Greater Poland Voivodeship
  - NZOZ Centrum Medyczne KERmed ( Site 2121), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz-Centrum Medyczne Pratia Bydgoszcz ( Site 2125), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 2159), Torun, Kuyavian-Pomeranian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca PAKS Małopolskie Centrum Sercowo-Naczyniowe ( Site 2141), Chrzanów, Lesser Poland Voivodeship
  - Maopolskie Centrum Kliniczne ( Site 2113), Krakow, Lesser Poland Voivodeship
  - Centrum Szybkiej Diagnostyki Kardiologicznej "Kardiomed" M. Żabówka E. Żabówka ( Site 2119), Tarnów, Lesser Poland Voivodeship
  - Private Practice - Dr. Robert Witek-Ośrodek Badań Klinicznych "METABOLICA" Lek. Robert Witek ( Site 2162), Tarnów, Lesser Poland Voivodeship
  - Beata Miklaszewicz & Dariusz Dabrowski CARDIAMED s.j. ( Site 2118), Legnica, Lower Silesian Voivodeship
  - NZOZ Twoja Przychodnia ( Site 2105), Lublin, Lublin Voivodeship
  - AMEDS CLINICAL RESEARCH ( Site 2166), Grodzisk Mazowiecki, Masovian Voivodeship
  - SPZOZ im. Jana Pawła II w Grodzisku Mazowieckim ( Site 2155), Grodzisk Mazowiecki, Masovian Voivodeship
  - Szpital Grochowski im. dr med. Rafała Masztaka SPZOZ ( Site 2139), Warsaw, Masovian Voivodeship
  - Narodowy Inst. Kardiologii Stefana kardynala Wyszynskiego-Inst. Badawczy.Centr.Wsparcia Badan Klinic ( Site 2132), Warsaw, Masovian Voivodeship
  - Centrum Medyczne Medyk ( Site 2101), Rzeszów, Podkarpackie Voivodeship
  - Trial Medica ( Site 2122), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 2148), Gdansk, Pomeranian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii Lek. med. Krzysztof Cymerman ( Site 2112), Gdynia, Pomeranian Voivodeship
  - Gabinet Kardiologiczno Internistyczny ( Site 2111), Gdynia, Pomeranian Voivodeship
  - NZOZ Sopockie Centrum Badan Kardiologicznych Pro Cordis Pawel Miekus ( Site 2130), Sopot, Pomeranian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca II Oddział Kardiologiczny ( Site 2140), Bielsko-Biala, Silesian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca ( Site 2145), Dąbrowa Górnicza, Silesian Voivodeship
  - Centrum Medyczne Pratia Katowice ( Site 2108), Katowice, Silesian Voivodeship
  - Clinical Medical Research ( Site 2102), Katowice, Silesian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca ( Site 2142), Tychy, Silesian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska dr n.med. Andrzej Tomasik ( Site 2146), Zabrze, Silesian Voivodeship
  - Poradnia Kardiologiczna KOS-Zawal ( Site 2104), Elblag, Warmian-Masurian Voivodeship
  - SOMED CR ( Site 2160), Lodz, Łódź Voivodeship
  - Instytut Centrum Zdrowia Matki Polki ( Site 2165), Lodz, Łódź Voivodeship
  - Velocity Skierniewice Sp. z o. o. ( Site 2114), Skierniewice, Łódź Voivodeship
  - Polsko Amerykanskie Kliniki Serca - Zgierskie ( Site 2144), Zgierz, Łódź Voivodeship
- Puerto Rico (4):
  - Clinical Research Investigator Group ( Site 3701), Bayamón
  - Investigadores del Este LLC ( Site 3700), Humacao
  - Ponce Medical School Foundation Inc. ( Site 3702), Ponce
  - Latin Clinical Trial Center ( Site 3704), San Juan
- South Africa (24):
  - Phoenix Pharma ( Site 2204), Port Elizabeth, Eastern Cape
  - IATROS INTERNATIONAL ( Site 2206), Bloemfontein, Free State
  - Lenasia Clinical Trial Centre - Johannesburg ( Site 2266), Johannesburg, Gauteng
  - Bara Cardiology Research ( Site 2258), Johannesburg, Gauteng
  - Helen Joseph Hospital-Clinical HIV Research Unit ( Site 2230), Johannesburg, Gauteng
  - Futurex Clinical. Dr Soraya Cassimjee INC ( Site 2269), Johannesburg, Gauteng
  - Netcare Sunninghill Hospital ( Site 2257), Johannesburg, Gauteng
  - Midrand Medical Centre ( Site 2202), Midrand, Gauteng
  - Zinakekele Medicall Centre ( Site 2225), Moloto, Gauteng
  - Clinical Trial Systems ( Site 2210), Pretoria, Gauteng
  - Sefako Makgatho Health Sciences University ( Site 2268), Pretoria, Gauteng
  - Jongaie Research ( Site 2211), Pretoria West, Gauteng
  - Wits Clinical Research ( Site 2220), Soweto, Gauteng
  - Enhancing Care Foundation-ECF research pharmacy ( Site 2213), Durban, KwaZulu-Natal
  - Private Practice - Dr. Neyaseelan Gounden ( Site 2207), Durban, KwaZulu-Natal
  - Tiervlei Trial Centre-Clinical ( Site 2205), Bellville, Cape Town, Western Cape
  - Helderberg Research Institute ( Site 2231), Cape Town, Western Cape
  - TREAD Research ( Site 2212), Cape Town, Western Cape
  - Excellentis Clinical Trial Consultants ( Site 2221), George, Western Cape
  - TASK Eden ( Site 2227), George, Western Cape
  - Be Part Yoluntu Centre ( Site 2209), Paarl, Western Cape
  - Paarl Research Centre ( Site 2214), Paarl, Western Cape
  - Tsitsikamma Clinical Research Initiative (TCRI) ( Site 2226), Plettenberg Bay, Western Cape
  - Clinical Projects Research ( Site 2265), Worcester, Western Cape
- South Korea (10):
  - Seoul National University Bundang Hospital ( Site 3005), Seongnam, Kyonggi-do
  - Ajou University Hospital ( Site 3006), Suwon, Kyonggi-do
  - Dong-A University Hospital ( Site 3013), Busan, Pusan-Kwangyokshi
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 3003), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 3001), Seoul
  - Kangbuk Samsung Hospital ( Site 3009), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 3002), Seoul
  - Asan Medical Center ( Site 3004), Seoul
  - Samsung Medical Center-cardiology ( Site 3000), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 3007), Seoul
- Spain (23):
  - Hospital Universitario de Torrevieja ( Site 2351), Torrevieja, Alicante
  - Hospital Universitario Reina Sofia-Medicina Interna ( Site 2362), Córdoba, Andalusia
  - Hospital Universitario Virgen de la Victoria-UGC Endocrinologia y nutricion ( Site 2323), Málaga, Andalusia
  - Hospital Universitario Virgen de Valme-Internal Medicine ( Site 2336), Seville, Andalusia
  - Corporació de Salut del Maresme i la Selva ( Site 2365), Calella, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 2342), Barcelona, Catalonia
  - EAP Osona Sud - Alt Congost S.L.P ( Site 2311), Centelles, Catalonia
  - Hospital Universitari de Bellvitge-Unitat de Lipids i Risc Vascular ( Site 2327), L'Hospitalet de Llobregat, Catalonia
  - CHUS - Hospital Clinico Universitario-Cardiology - Clinical Research Unit ( Site 2320), Santiago de Compostela, La Coruna
  - Complejo Asistencial Universitario de León - Hospital de León ( Site 2339), León, Leon
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-Endocrinologia y Nutrición ( Site 2344), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Fundacion ALcorcon ( Site 2353), Alcorcón, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal ( Site 2337), Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz ( Site 2333), Madrid, Madrid, Comunidad de
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA ( Site 2348), Majadahonda, Madrid, Comunidad de
  - Hospital Clínico Universitario Virgen de la Arrixaca-CARDIOLOGÍA ( Site 2328), El Palmar, Murcia, Murcia, Region de
  - Vithas Hospital Sevilla-Unidad de Salud Metabólica. Diabetes y Obesidad ( Site 2349), Castilleja de la Cuesta, Sevilla
  - Hospital Universitari i Politecnic La Fe ( Site 2340), Valencia, Valencia
  - HOSPITAL CLINICO DE VALENCIA-CARDIOLOGY ( Site 2321), Valencia, Valenciana, Comunitat
  - Hospital La Luz ( Site 2366), Madrid
  - Hospital La Princesa ( Site 2334), Madrid
  - Hospital Clinico San Carlos-Cardiology ( Site 2325), Madrid
  - Hospital Universitari Joan XXIII de Tarragona ( Site 2350), Tarragona
- Taiwan (10):
  - Mackay Memorial Hospital -Tamsui Branch ( Site 3108), New Taipei City, New Taipei
  - Chi Mei Medical Center-Cardiology ( Site 3104), Tainan, Tainan
  - Changhua Christian Hospital ( Site 3101), Changhua
  - Kaohsiung Medical University Hospital ( Site 3109), Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3102), Kaohsiung City
  - China Medical University Hospital ( Site 3103), Taichung
  - National Taiwan University Hospital ( Site 3100), Taipei
  - Taipei Medical University Hospital-Cardiology ( Site 3107), Taipei
  - Taipei Veterans General Hospital ( Site 3106), Taipei
  - Tri-Service General Hospital ( Site 3110), Taipei
- Turkey (Türkiye) (17):
  - Hacettepe Universite Hastaneleri ( Site 2500), Altindağ, Ankara
  - Ege Universitesi Hastanesi-Cardilogy Department ( Site 2502), Bornova, İzmir
  - I.E.U. Medical Point Hastanesi ( Site 2521), Cordaleo, İzmir
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri-endocrine ( Site 2522), Melikgazi, Kayseri
  - Adana Sehir Egitim ve Arastirma Hastanesi ( Site 2511), Adana
  - SBÜ GÜLHANE EĞİTİM VE ARAŞTIRMA HASTANESİ ( Site 2524), Ankara
  - Ankara Bilkent Şehir Hastanesi-cardiology ( Site 2501), Ankara
  - Antalya Egitim ve Arastırma Hastanesi-Cardiology ( Site 2518), Antalya
  - Çanakkale Onsekiz Mart Üniversitesi ( Site 2509), Çanakkale
  - Trakya University ( Site 2523), Edirne
  - Eskisehir Osmangazi University-Cardiology ( Site 2510), Eskişehir
  - Istanbul University Cerrahpasa Medical School Internal Diseases Institute ( Site 2528), Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi ( Site 2520), Istanbul
  - Kocaeli Üniversitesi-Cardiology ( Site 2516), Kocaeli
  - NECMETTIN ERBAKAN MERAM MEDICAL FAC.-cardiology ( Site 2513), Konya
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi ( Site 2525), Malatya
  - Ondokuz Mayis Universitesi Saglik Uygulama ve Arastirma Merkezi ( Site 2527), Samsun
- United Kingdom (12):
  - West Walk Surgery ( Site 2602), Bristol, Bristol, City of
  - Velocity Clinical Research Romford ( Site 2615), Bristol, Bristol, City of
  - Royal Devon & Exeter Hospital-Patient Recruitment Centre: Exeter ( Site 2605), Exeter, Devon
  - Walsall Manor Hospital ( Site 2600), Walsall, Devon
  - Barts Health NHS Trust-William Harvey Clinical Research Centre ( Site 2603), London, England
  - NIHR Commercial Recruitment Delivery Centre: Newcastle ( Site 2606), Newcastle upon Tyne, England
  - Golden Jubilee National Hospital ( Site 2613), Clydebank, Glasgow City
  - Velocity Clinical Research Romford ( Site 2618), Romford, London, City of
  - Lakeside Surgery ( Site 2601), Corby, Northamptonshire
  - Velocity Clinical Research, Leicester ( Site 2614), Leicester
  - Manchester Royal Infirmary ( Site 2612), Manchester
  - Northern General Hospital ( Site 2611), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26301&tenant=MT_MSD_9011